CLINICAL TRIAL: NCT00426270
Title: Clinical Study to Evaluate the Efficacy and Safety of Octagam® 10% in Idiopathic Thrombocytopenic Purpura in Adults
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Octagam 10% in Idiopathic Thrombocytopenic Purpura in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAM10-02
Record Dates: First submitted 2007-01-22; First posted 2007-01-24 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Octagam 10% 1 g/kg/day (Experimental): Participants received Octagam 10% (human normal immunoglobulin) 1 g/kg intravenously once a day for 2 days.
  Interventions: Drug: Octagam 10%

INTERVENTIONS:
Drug: Octagam 10% — Octagam 10% was supplied as a ready-to-use solution in glass bottles.
  Other Names: Human normal immunoglobulin

SUMMARY:
Octagam is a solvent/detergent-treated human normal immunoglobulin (IGIV) solution for intravenous administration. Octagam 5% is currently registered in about 80 countries. This study evaluated the efficacy and safety of Octagam 10% in Idiopathic Thrombocytopenic Purpura (ITP) in adults. As Octagam 10% is essentially similar to Octagam 5%, it is expected that Octagam 10% is as efficacious and safe (in respect to viral safety) as Octagam 5%.

DETAILED DESCRIPTION:
The primary objective of the study was to investigate the efficacy of Octagam® 10% in correcting platelet count. The blood count as well as laboratory chemistry were checked repeatedly up to day 21.

The secondary objective of the study was to investigate the safety of Octagam® 10%. Safety was assessed by monitoring vital signs, evaluating adverse events, assessing laboratory parameters, and by viral safety testing.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of Idiopathic Thrombocytopenic Purpura (ITP) according to standard criteria.
* Platelet count ≤ 20 x 10^9/L.

Key Exclusion Criteria:

* Chronic refractory ITP patients.
* Thrombocytopenia secondary to other diseases, or drug related thrombocytopenia.
* Administration of IGIV, anti-D, or other platelet enhancing drugs within 30 days before enrollment.
* Administration of thrombocyte concentrates within 72 hours before baseline.
* Experimental treatment (eg, rituximab) within 3 months before enrollment.
* Prophylactic preoperative treatment for elective splenectomy.
* Severe liver or kidney disease.
* Pregnant or nursing female.
* History of hypersensitivity to blood or plasma derived products.
* Emergency operation.
* Live viral vaccination within the last month prior to study entry.
* Known IgA deficiency and antibodies against IgA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, MD, Study Director — Octapharma
Locations (1):
- Contact Octapharma for information, Vienna, Austria

REFERENCES:
- [Derived] Robak T, Mainau C, Pyringer B, Chojnowski K, Warzocha K, Dmoszynska A, Straub J, Imbach P. Efficacy and safety of a new intravenous immunoglobulin 10% formulation (octagam(R) 10%) in patients with immune thrombocytopenia. Hematology. 2010 Oct;15(5):351-9. doi: 10.1179/102453310X12719010991867. PMID 20863431

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was incorrectly enrolled in the study and was not included in the efficacy analyses but was included in the safety population.
Period: Overall Study
Arm/Group | Octagam 10% 1 g/kg/Day
Started | 116
Completed | 110
Not Completed | 6
Not completed — Incorrectly Enrolled in the Study | 1
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received at least 1 dose of study medication.
Arm/Group | Octagam 10% 1 g/kg/Day
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (19.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Clinical Response
Description: A clinical response is defined as an increase in platelet count to ≥ 50*10^9/L on any day from Day 2 to Day 7.
Time Frame: Day 2 to Day 7
Population: Full analysis set: All participants who received at least 1 dose of study medication, satisfied all major entry criteria, and had at least 1 post-baseline measurement of platelet count.
Measure: Number; unit: Percentage of participants
Arm/Group | Octagam 10% 1 g/kg/Day
Number analyzed (Participants) | 115
Percentage of participants | 80.0

2. Secondary Outcome: Time to Achieve a Clinical Response
Description: A clinical response is defined as an increase in platelet count to ≥ 50*10^9/L on any day from Day 2 to Day 7.
Time Frame: Day 2 to Day 7
Population: Full analysis set: All participants who received at least 1 dose of study medication, satisfied all major entry criteria, and had at least 1 post-baseline measurement of platelet count. Only participants with a clinical response were included in the analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Octagam 10% 1 g/kg/Day
Number analyzed (Participants) | 92
Days | 2.1 (1.08)

3. Secondary Outcome: Maximum Platelet Count
Description: Platelet count was assessed on Days 2 through 7 and on Days 14, 21, and 63. The maximum measured platelet count is reported.
Time Frame: Day 2 to the end of the study (Day 63)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: *10^9/L
Arm/Group | Octagam 10% 1 g/kg/Day
Number analyzed (Participants) | 115
*10^9/L | 221.6 (142.66)

4. Secondary Outcome: Duration of the Clinical Response
Description: The duration of the clinical response was the number of days that the platelet count remained ≥ 50*10^9/L. Platelet count was assessed on Days 2 through 7 and on Days 14, 21, and 63. A conservative method was used to calculate the duration of the clinical response. For example, if the platelet count was ≥ 50*10^9/L on Day 7 and dropped below 50*10^9/L at Day 14, Day 7 was used as the last day to calculate the duration of the clinical response. The same procedure was used if the platelet count dropped below 50*10^9/L at Day 21 from Day 14 or Day 63 from Day 21.
Time Frame: Day 2 to the end of the study (Day 63)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Octagam 10% 1 g/kg/Day
Number analyzed (Participants) | 92
Days | 24.1 (23.88)

5. Secondary Outcome: Percentage of Participants With None, Minor, Mild, or Moderate Bleeding at Day 7
Description: The investigator evaluated the severity of bleeding using the following rating scale: None (definitely no haemorrhage of any kind), Minor (few petechiae [≤ 100 total] and/or ≤ 5 small bruises [≤ 3 cm diameter], no mucosal bleeding), Mild (many petechiae [> 100 total] and/or > 5 large bruises [> 3 cm diameter], no mucosal bleeding), Moderate (overt mucosal bleeding [epistaxis, gum bleeding, oropharyngeal blood blisters, menorrhagia, gastrointestinal bleeding, etc] that does not require immediate medical attention or intervention).
Time Frame: Day 7
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Octagam 10% 1 g/kg/Day
Number analyzed (Participants) | 115
Percentage of participants
  None | 80.9
  Minor | 13.0
  Mild | 2.6
  Moderate | 0.9
  Missing | 2.6

ADVERSE EVENTS:
Description: Safety population: All participants who received at least 1 dose of study medication.
Arm/Group | Octagam 10% 1 g/kg/Day
Serious Adverse Events (participants affected / at risk) | 14/116
Other Adverse Events (participants affected / at risk) | 79/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octagam 10% 1 g/kg/Day (N=116)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Extradural haematoma (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Octagam 10% 1 g/kg/Day (N=116)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 6
Nausea (Gastrointestinal disorders) | 7
Pyrexia (General disorders) | 21
Heart rate decreased (Investigations) | 18
Heart rate increased (Investigations) | 25
Headache (Nervous system disorders) | 35
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No